CLINICAL TRIAL: NCT00572208
Title: Gabapentin for Postoperative Pain Management After Cardiac Surgery With Median Sternotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Vibeke Hjortdal, Professor, Consultant, Dr. Sci., PhD., Cardiothoracic and Vascular Surgery Department, Aarhus University Hospital, Skejby
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gabapentin01; 2007-001479-12
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Gabapentin group
  Interventions: Drug: Gabapentin group
- 2 (No Intervention): placebo

INTERVENTIONS:
Drug: Gabapentin group — Gabapentin group:
  Preoperative (2 h before surgery): Tablet Gabapentin 1200 mg (blinded)
  1. st Postoperative day: Tablet Gabapentin 300 mg twice a day (blinded)
  2. nd Postoperative day: Tablet Gabapentin 300 mg twice a day (blinded)
  3. rd Postoperative day: Tablet Gabapentin 300 mg twice a day (blinded)
  4. th Postoperative day: Tablet Gabapentin 300 mg twice a day (blinded)
  5. th Postoperative day: Tablet Gabapentin 300 mg twice a day (blinded)
  Arms: 1

SUMMARY:
In this study we will focus on the postoperative recovery. A successful postoperative recovery should bring the patient to at least to the pre-surgical level. This can probably be achieved by a multimodal approach where at least postoperative pain and PONV are managed.

The surgical injury results in immobilisation which again can result in impaired cardiac, respiratory and musculoskeletal system. Pain relief is a prerequisite for mobilisation and an early return to the pre-surgical level. The preferred drugs for postoperative pain management are opioids. Although opioids are known to be an effective analgesia, they have a series of side effects: nausea, vomiting, constipation, respiratory deficiency, delirium among others.

Gabapentin has been tested for post operative pain. Randomized Clinical Trials have reported a significant better pain scores with Gabapentin in several studies -most of them restricted to the postoperative period in the post-anaesthesia care unit in many different kind of surgeries.

We want to test if Gabapentin can be used instead of opioids for treatment of postoperative pain after heart surgery by median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective cardiac surgery with median sternotomy at the department of cardiac surgery, Aarhus University Hospital, Skejby.
2. Patients older than 18 years.

Exclusion Criteria:

1. Patients unable to cooperate.
2. Known allergy for Gabapentin or opioids.
3. Acute pancreatitis
4. History of gastric or peptic ulcer.
5. History of alcohol or drug abuse.
6. Chronic pain or daily intake of analgesics or corticosteroids.
7. Gastrointestinal obstruction
8. Impaired liver function.
9. Impaired kidney function.
10. Previous operation with median sternotomy
11. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Pain | 1 month
Morphine consumption | 1 month

SECONDARY OUTCOMES:
PONV | 1 month
Medication side effects | 1 month
Hospital stay | 1 month
VAS score and medication 30 days after the operation | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Hjortdal, MD, Dr.sci, Principal Investigator — Cardiothoracic and Vascular Surgery Department, Aarhus University Hospital, Skejby
Locations (2):
- Denmark (2):
  - Cardiothoracic and Vascular Surgery Department, Aarhus University Hospital, Skejby, Aarhus
  - Cardiothoracic and vascular department, Skejby Sygehus, Aarhus